CLINICAL TRIAL: NCT01915303
Title: A Phase II Trial to Assess the Efficacy and Safety of Pasireotide s.c. Alone or in Combination With Cabergoline in Patients With Cushing's Disease
Brief Title: Study of the Efficacy and Safety of Pasireotide s.c. +/- Cabergoline in Patients With Cushing's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230B2411
Record Dates: First submitted 2013-06-10; First posted 2013-08-02 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-08

CONDITIONS: Cushings Disease
Keywords: pituitary tumors; pasireotide; cabergoline; combination treatment; UFC; hormone disorder; cortisol; adrenocorticotropic hormone; Cushing Disease
MeSH Terms: conditions — Adrenocortical Hyperfunction; Pituitary Neoplasms; Pituitary ACTH Hypersecretion | interventions — pasireotide; Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- pasireotide +/- cabergoline (Experimental): pasireotide alone or with cabergoline
  Interventions: Drug: Pasireotide with or without cabergoline

INTERVENTIONS:
Drug: Pasireotide with or without cabergoline — The trial consisted of Pasireotide-untreated patients who started pasireotide 0.6mg twice a day for 8 weeks. If biochemical control was not achieved by the end of the 8 weeks, and the 0.6mg dose is well-tolerated, the dose was increased to 0.9mg twice a day for another 8 weeks. If biochemical control is not achieved, cabergoline was added and patients began combination treatment with cabergoline at the starting dose of 0.5mg once a day for 8 weeks. If biochemical control is still not achieved at the end of the third 8 week period, the dose of cabergoline was increased to 1.0mg once a day. Patients could also immediately start the combination treatment by adding cabergoline 0.5mg once a day at study entry to their current maximal tolerated dose of pasireotide. Patients continued with the combination treatment for 8 weeks. If biochemical control was not not achieved by the end of the 8 week period, the dose of cabergoline was increased to 1mg once a day.

SUMMARY:
The main purpose of this prospective, multicenter, open-label phase II study, was to evaluate the efficacy and safety of pasireotide alone or in combination with cabergoline in patients with Cushing's disease.

DETAILED DESCRIPTION:
This was an open-label, multi-center, international, non-comparative study with adult patients with confirmed diagnosis of Cushing's disease. Given the fact that CD patients may need a multimodality treatment approach, the trial design aimed to mimic CD treatment by using a medical stepwise approach. Therefore, the whole patient population started treatment with Pasireotide and only in patients within this population who did not achieve biochemical control, cabergoline was added.

The whole patient population had never received pasireotide or had received it in the past (reasons of discontinuation not related to safety).

Core Phase

* Pasireotide naïve patients started pasireotide monotherapy at the dose of 0.6 mg s.c. bid. If at the end of the 8 week treatment period, the biochemical control was not achieved and the 0.6mg bid dose was well tolerated, the pasireotide dose was increased to 0.9mg bid. If the 0.9mg bid dose of pasireotide did not lead to biochemical control, cabergoline was added with a starting dose of 0.5mg qd. If the combination dose of 0.9mg bid of pasireotide plus 0.5mg qd cabergolinedid not achieve biochemical control, the cabergoline dose will be increased to 1.0mg qd.
* Patients who were currently being treated with maximal tolerated doses of pasireotide monotherapy for at least 8 weeks at screening without achieving normal mUFC, entered the study with a combination therapy starting with cabergoline 0.5mg qd.

Extension Phase

• After 35 weeks of treatment in core phase, patients had the option to continue study treatment if pasireotide was not yet approved for commercial use and/or reimbursed - if country reimbursement was applicable - in each respective country, or until 31st December 2017, or once an applicable roll over protocol became available, or whichever occurred first.

Novartis had a local transition plan in order to ensure that all trial patients had access to the study medication without any delay in their treatment

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent obtained prior to screening procedures
2. Adult patients with confirmed diagnosis of ACTH-dependent Cushing's disease as evidenced by all of the following:

   1. The mean of three 24-hour urine samples collected within 2 weeks > 1xULN with 2 out of 3 samples >ULN
   2. Morning plasma ACTH within the normal or above normal range
   3. Either MRI confirmation of pituitary adenoma > 6 mm, or inferior petrosal sinus gradient >3 after CRH stimulation for those patients with a tumor less than or equal to 6 mm*. For patients who have had prior pituitary surgery, histopathology confirming an ACTH staining adenoma *If IPSS had previously been performed without CRH (e.g. with DDAVP), then a central to peripheral pre-stimulation gradient > 2 was required. If IPSS had not previously been performed, IPSS with CRH stimulation was required.
3. Patients with de novo Cushing's disease could only be included only if they were not considered candidates for pituitary surgery (e.g. poor surgical candidates, surgically unapproachable tumors, patients who refused to have surgical treatment)
4. Male or female patients aged 18 years or greater
5. Karnofsky performance status ≥ 60 (i.e. required occasional assistance, but was able to care for most of their personal needs)
6. Patients on medical treatment for Cushing's disease the following washout periods must have been completed before screening assessments were performed

   * Inhibitors of steroidogenesis (ketoconazole, metyrapone): 1 week
   * Pituitary directed agents: Dopamine agonists (bromocriptine, cabergoline) and PPARγ agonists (rosiglitazone or pioglitazone): 4 weeks
   * Octreotide LAR, Lanreotide SR and Lanreotide autogel: 14 weeks
   * Octreotide (immediate release formulation): 1 week
   * Progesterone receptor antagonist (mifepristone): 4 weeks
7. Patients could have been considered to enter the trial if they met any one of the following criteria: 1) They were naive to pasireotide 2) They had received pasireotide in the past and have been discontinued because of lack of efficacy (2 weeks for washout prior to screening for patients treated with pasireotide subcutaneously and 12 weeks of washout prior to screening for patients treated with pasireotide LAR) 3) Patients who were on maximal tolerated dose but had not achieved biochemical control
8. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, if they were using highly effective methods of contraception during dosing and for 30 days after stopping study medication.
9. Male participants in the trial must have agreed to use a condom during intercourse, and not to father a child during the study and for the period of 30 days following stopping of the study treatment.

Exclusion criteria:

1. Patients with compression of the optic chiasm that caused any visual field defect that required surgical intervention
2. Diabetic patients with poor glycemic control as evidenced by HbA1c >8%
3. Patients with risk factors for torsade de pointes, i.e. patients with a baseline QTcF >450 ms in males, and > 460 ms in females. hypokalemia, hypomagnesaemia, uncontrolled hypothyroidism, family history of long QT syndrome, or concomitant medications known to prolong QT interval.
4. Patients with clinically significant valvular disease.
5. Patients with Cushing's syndrome due to ectopic ACTH secretion
6. Patients with hypercortisolism secondary to adrenal tumors or nodular (primary) bilateral adrenal hyperplasia
7. Patients who had congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, advanced heart block, history of acute MI less than one year prior to study entry or clinically significant impairment in cardiovascular function
8. Patients with liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis, or patients with ALT/AST > 2 X ULN, serum bilirubin >2.0 X ULN
9. Patients with serum creatinine >2.0 X ULN
10. Patients with WBC <3 X 10e9/L; Hb 90% < LLN; PLT <100 X 10e9/L
11. Patients with presence of Hepatitis B surface antigen (HbsAg)
12. Patients with presence of Hepatitis C antibody test (anti-HCV)
13. Patients with severe hepatic impairment (Child Pugh C) and hypersensitivity to pasireotide or cabergoline
14. Patients with lung, pericardial, and retroperitoneal fibrosis; gastro-duodenal ulcer or digestive haemorrhage, galactose intolerance, Parkinson's disease, uncontrolled hypertension and Raynauds syndrome.
15. Pregnant or nursing (lactating) women where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/ml)
16. Patients with end-stage renal failure and/or hemodialysis
17. Patients with presence of active or suspected acute or chronic uncontrolled infection
18. Patients with a history of non-complance to medical regimens or who were considered potentially unreliable or were unable to complete the entire study
19. Patients with presence of Hepatitis B surface antigen (HbsAg)
20. Patients with presence of Hepatitis C antibody test (anti-HCV)
21. Patients with severe hepatic impairment (Child Pugh C) and hpersensitivity to pasireotide or cabergoline
22. Patients with lung, pericardial, and retroperitoneal fibrosis; gastroduodenal ulcer or digestive haemorrhage, galactose intolerance, Parkinson's disease, uncontrolled hypertension and Raynaud's syndrome
23. Pregnant or nursing (lactating) women where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5mIU/mL)
24. Patients with end-stage renal failure and/or hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2016-09-05 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (2):
  - University of Alabama at Birmingham The Kirklin Clinic, Birmingham, Alabama
  - Oregon Health and Science University SOM230B2411, Portland, Oregon
- Novartis Investigative Site, Caba, Buenos Aires, Argentina
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Brazil (4):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Bogota, Cundinamarca, Colombia
- Novartis Investigative Site, Vandœuvre-lès-Nancy, France
- Novartis Investigative Site, Erlangen, Germany
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Budapest, Hungary
- India (3):
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Chandigarh
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Napoli, Italy
- Novartis Investigative Site, Wilayah Persekutuan, Malaysia
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Durango
- Novartis Investigative Site, Rotterdam, Netherlands
- Spain (2):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Alzira, Valencia
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Pendik / Istanbul, Turkey
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Feelders RA, Fleseriu M, Kadioglu P, Bex M, Gonzalez-Devia D, Boguszewski CL, Yavuz DG, Patino H, Pedroncelli AM, Maamari R, Chattopadhyay A, Biller BMK, Pivonello R. Long-term efficacy and safety of subcutaneous pasireotide alone or in combination with cabergoline in Cushing's disease. Front Endocrinol (Lausanne). 2023 Oct 9;14:1165681. doi: 10.3389/fendo.2023.1165681. eCollection 2023. PMID 37876540

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Pasireotide montherapy (0.6 mg bid to 0.9 mg bid) was administered until the biochemical control was achieved and if not achieved, a combination was administered: pasireotide (0.9 mg bid) + cabergoline (0.5 QD to 1 mg QD). Patients were able to add cabergoline at anytime during core and extension
Period: Core Phase
Arm/Group | All Patients
Started | 68
Completed | 52
Not Completed | 16
Not completed — Adverse Event | 7
Not completed — Unsatisfactory therapeutic effect | 3
Not completed — Death | 2
Not completed — Protocol Violation | 2
Not completed — Abnormal lab value | 1
Not completed — Withdrawal by Subject | 1
Period: Extension Phase
Arm/Group | All Patients
Started | 29
Completed | 12
Not Completed | 17
Not completed — Unsatisfactory therapeutic effect | 8
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 3
Not completed — Death | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 68
Age, Customized [Number; unit: participants]
  < 65 years | 64
  ≥ 65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 44
  Asian | 9
  Native American | 5
  Black | 2
  Other | 8
Cushing's disease status [Number; unit: Participants] — De novo = newly diagnosed and persistent/recurrent = xxxxxxxx
  Participants
    De novo | 10
    Persistent/recurrent | 58
Clinical symptoms of facial rubor [Number; unit: Participants] — Clinical symptoms of CD for facial rubor by severity
  Participants
    None | 10
    Mild | 17
    Moderate | 11
    Severe | 4
    Not done | 26
Clinical symptoms of hirsutism [Number; unit: Participants] — Clinical symptoms of CD for hirsutism by severity
  Participants
    None | 13
    Mild | 12
    Moderate | 7
    Severe | 3
    Not done | 33
Clinical symptoms of striae [Number; unit: Participants] — Clinical symptoms of CD for striae by severity
  Participants
    None | 20
    Mild | 10
    Moderate | 4
    Severe | 8
    Not done | 26
Clinical symptoms of supraclavicular fat pad [Number; unit: Participants] — Clinical symptoms of CD for supraclavicular fat pad by severity
  Participants
    None | 8
    Mild | 17
    Moderate | 13
    Severe | 4
    Not done | 26
Clinical symptoms of dorsal fat pad [Number; unit: Participants] — Clinical symptoms of CD for dorsal fat pad severity
  Participants
    None | 3
    Mild | 19
    Moderate | 14
    Severe | 6
    Not done | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders With Mean Urinary Free Cortisol (mUFC) ≤ 1.0xULN Collected or Imputed at Week 35
Description: Participants who attained mUFC ≤ 1.0 x ULN (upper limit of normal) with pasireotide alone or in combination with cabergoline. The 24h-UFC concentration results from three samples, collected during the screening period, were averaged to obtain the Baseline urinary free cortisol level. mean 24h-UFC was determined from two 24-hour urine collections collected on two consecutive days that occurred before the visit. Imputation: subjects who completed the end of treatment visit at Week 35, but had missing evaluation of mean urinary free cortisol (mUFC). The last available mUFC assessment at or after previous visit (week) before last week was carried forward as the last week mUFC assessment.
Time Frame: Baseline up to week 35
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | All Patients
Number analyzed (Participants) | 68
percentage of responders | 50.0 [37.6 to 62.4]

2. Secondary Outcome: Mean Urinary Free Cortisol (mUFC) at Scheduled Visits
Description: Mean value of mUFC at each scheduled visit was determined from two 24-hour urine collections collected on two consecutive days that occurred before the visit when UFC was measured.
Time Frame: Baseline, weeks 2, 4, every 4 or 5 weeks during core, every 8 weeks during extension
Population: Full analysis set. The data beyond Week 139 should be interpreted with caution given that small number of subjects were monitored
Measure: Mean (Standard Deviation); unit: nmol/24h
Arm/Group | All Patients
Number analyzed (Participants) | 68
nmol/24h
  Baseline | 501.6 (488.66)
  Core Week 2 n-8: number analyzed (Participants) | 8
  Core Week 2 n-8 | 217.0 (100.69)
  Core Week 4 n=59: number analyzed (Participants) | 59
  Core Week 4 n=59 | 242.1 (203.47)
  Core Week 8 n=58: number analyzed (Participants) | 58
  Core Week 8 n=58 | 230.0 (195.21)
  Core Week 13 n=51: number analyzed (Participants) | 51
  Core Week 13 n=51 | 231.0 (240.98)
  Core Week 17 n=57: number analyzed (Participants) | 57
  Core Week 17 n=57 | 310.3 (429.64)
  Core Week 22 n=50: number analyzed (Participants) | 50
  Core Week 22 n=50 | 214.0 (202.80)
  Core Week 26 n=54: number analyzed (Participants) | 54
  Core Week 26 n=54 | 211.6 (173.58)
  Core Week 31 n=46: number analyzed (Participants) | 46
  Core Week 31 n=46 | 154.3 (104.16)
  Core Week 35 n=45: number analyzed (Participants) | 45
  Core Week 35 n=45 | 184.8 (140.13)
  Ext Week 43 n=22: number analyzed (Participants) | 22
  Ext Week 43 n=22 | 136.1 (91.13)
  Ext Week 51 n=20: number analyzed (Participants) | 20
  Ext Week 51 n=20 | 156.8 (108.91)
  Ext Week 59 n=24: number analyzed (Participants) | 24
  Ext Week 59 n=24 | 157.7 (111.63)
  Ext Week 67 n=17: number analyzed (Participants) | 17
  Ext Week 67 n=17 | 213.8 (194.99)
  Ext Week 75 n=18: number analyzed (Participants) | 18
  Ext Week 75 n=18 | 157.6 (166.28)
  Ext Week 83 n=20: number analyzed (Participants) | 20
  Ext Week 83 n=20 | 157.9 (134.98)
  Ext Week 91 n=18: number analyzed (Participants) | 18
  Ext Week 91 n=18 | 180.0 (302.36)
  Ext Week 99 n=13: number analyzed (Participants) | 13
  Ext Week 99 n=13 | 222.5 (375.67)
  Ext Week 107 n=12: number analyzed (Participants) | 12
  Ext Week 107 n=12 | 118.5 (122.01)
  Ext Week 115 n=13: number analyzed (Participants) | 13
  Ext Week 115 n=13 | 126.0 (80.09)
  Ext Week 123 n=13: number analyzed (Participants) | 13
  Ext Week 123 n=13 | 147.5 (157.77)
  Ext Week 131 n=11: number analyzed (Participants) | 11
  Ext Week 131 n=11 | 76.4 (49.92)
  Ext Week 139 n=9: number analyzed (Participants) | 9
  Ext Week 139 n=9 | 92.9 (73.18)
  Ext Week 147 n=9: number analyzed (Participants) | 9
  Ext Week 147 n=9 | 90.1 (55.31)
  Ext Week 155 n=4: number analyzed (Participants) | 4
  Ext Week 155 n=4 | 76.3 (39.05)
  Ext Week 163 n=6: number analyzed (Participants) | 6
  Ext Week 163 n=6 | 141.1 (142.42)
  Ext Week 171 n=6: number analyzed (Participants) | 6
  Ext Week 171 n=6 | 89.5 (61.87)
  Ext Week 179 n=4: number analyzed (Participants) | 4
  Ext Week 179 n=4 | 61.3 (43.06)
  Ext Week 187 n=4: number analyzed (Participants) | 4
  Ext Week 187 n=4 | 89.9 (52.44)
  Ext Week 195 n=3: number analyzed (Participants) | 3
  Ext Week 195 n=3 | 46.1 (40.21)
  Ext Week 203 n=4: number analyzed (Participants) | 4
  Ext Week 203 n=4 | 194.0 (259.15)
  Ext Week 211 n=3: number analyzed (Participants) | 3
  Ext Week 211 n=3 | 107.3 (37.68)
  Ext Week 219 n=2: number analyzed (Participants) | 2
  Ext Week 219 n=2 | 70.6 (46.74)
  Ext Week 227 n=2: number analyzed (Participants) | 2
  Ext Week 227 n=2 | 47.1 (7.99)
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 62.0 (23.83)
  Ext Week 243 n=1: number analyzed (Participants) | 1
  Ext Week 243 n=1 | 117.7
  Ext Week 251 n=1: number analyzed (Participants) | 1
  Ext Week 251 n=1 | 202.9
  Ext Week 267 n=1: number analyzed (Participants) | 1
  Ext Week 267 n=1 | 249.0

3. Secondary Outcome: Percentage of Responders With Mean Urinary Free Cortisol (mUFC) ≤ 1.0xULN
Description: Actual mean value of mUFC at each scheduled visit was determined from two 24-hour urine collections collected on two consecutive days that occurred before the visit when UFC was measured.
Time Frame: Baseline up to week 235
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | All Patients
Number analyzed (Participants) | 68
percentage of responders
  Baseline | 4.4 [0.9 to 12.4]
  Core Week 17 n=57: number analyzed (Participants) | 57
  Core Week 17 n=57 | 28.1 [17.0 to 41.5]
  Core Week 35 n=45: number analyzed (Participants) | 45
  Core Week 35 n=45 | 48.9 [33.7 to 64.2]
  Ext Week 43 n=22: number analyzed (Participants) | 22
  Ext Week 43 n=22 | 63.6 [40.7 to 82.8]
  Ext Week 67 n=17: number analyzed (Participants) | 17
  Ext Week 67 n=17 | 47.1 [23.0 to 72.2]
  Ext Week 91 n=18: number analyzed (Participants) | 18
  Ext Week 91 n=18 | 61.1 [35.7 to 82.7]
  Ext Week 115 n=13: number analyzed (Participants) | 13
  Ext Week 115 n=13 | 76.9 [46.2 to 95.0]
  Ext Week 139 n=9: number analyzed (Participants) | 9
  Ext Week 139 n=9 | 77.8 [40.0 to 97.2]
  Ext Week 163 n=6: number analyzed (Participants) | 6
  Ext Week 163 n=6 | 66.7 [22.3 to 95.7]
  Ext Week 187 n=4: number analyzed (Participants) | 4
  Ext Week 187 n=4 | 75.0 [19.4 to 99.4]
  Ext Week 211 n=3: number analyzed (Participants) | 3
  Ext Week 211 n=3 | 66.7 [9.4 to 99.2]
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 100 [29.2 to 100.0]

4. Secondary Outcome: Percentage of Participants Who Attain mUFC ≤ 1.0 x ULN or Have at Least 50% Reduction From Baseline in mUFC
Description: as for outcome 3
Time Frame: Baseline up to week 235
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | All Patients
Number analyzed (Participants) | 68
percentage of responders
  Baseline | 4.4 [0.9 to 12.4]
  Core Week 17 n=57: number analyzed (Participants) | 57
  Core Week 17 n=57 | 54.4 [40.7 to 67.6]
  Core Week 35 n=45: number analyzed (Participants) | 45
  Core Week 35 n=45 | 68.9 [53.4 to 81.8]
  Ext Week 43 n=22: number analyzed (Participants) | 22
  Ext Week 43 n=22 | 86.4 [65.1 to 97.1]
  Ext Week 67 n=17: number analyzed (Participants) | 17
  Ext Week 67 n=17 | 76.5 [50.1 to 93.2]
  Ext Week 91 n=18: number analyzed (Participants) | 18
  Ext Week 91 n=18 | 83.3 [58.6 to 96.4]
  Ext Week 115 n=13: number analyzed (Participants) | 13
  Ext Week 115 n=13 | 92.3 [64.0 to 99.8]
  Ext Week 139 n=9: number analyzed (Participants) | 9
  Ext Week 139 n=9 | 77.8 [40.0 to 97.2]
  Ext Week 163 n=6: number analyzed (Participants) | 6
  Ext Week 163 n=6 | 83.3 [35.9 to 99.6]
  Ext Week 187 n=4: number analyzed (Participants) | 4
  Ext Week 187 n=4 | 100 [39.8 to 100.0]
  Ext Week 211 n=3: number analyzed (Participants) | 3
  Ext Week 211 n=3 | 66.7 [9.4 to 99.2]
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 100 [29.2 to 100.0]

5. Secondary Outcome: Duration (Weeks) of Controlled or Partially Controlled Response
Description: Duration of controlled or partially controlled response is defined as the period starting from the date of patient's first normalization (mUFC ≤ 1.0 x ULN) or at least 50% reduction from baseline up to the date when the patient's mUFC > 1.0 x ULN and the reduction from baseline falls to less than 50% from the first time
Time Frame: from the date patient's first normalization (mUFC ≤ 1.0xULN) or at least 50% reduction from baseline up to the date when the patient's mUFC > 1.0 x ULN
Population: Core and extension full analysis set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | All Patients
Number analyzed (Participants) | 68
weeks
  Core n=36: number analyzed (Participants) | 36
  Core n=36 | 13.1 [9.3 to 22.4]
  Extension n=20: number analyzed (Participants) | 20
  Extension n=20 | 22.0 [8.1 to 70.1]

6. Secondary Outcome: Plasma Adrenocorticotropic Hormone (ACTH)
Description: A pre-dose blood draw for plasma ACTH sampling was taken at visits. Samples were analyzed by a central laboratory.
Time Frame: Baseline, weeks 2, 4, every 4 or 5 weeks during core, every 8 weeks during extension
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | All Patients
Number analyzed (Participants) | 68
pmol/L
  Baseline | 16.3 (16.3)
  Core Week 2 n-62: number analyzed (Participants) | 62
  Core Week 2 n-62 | 12.4 (9.91)
  Core Week 4 n=63: number analyzed (Participants) | 63
  Core Week 4 n=63 | 14.2 (12.50)
  Core Week 8 n=61: number analyzed (Participants) | 61
  Core Week 8 n=61 | 13.3 (11.90)
  Core Week 13 n=53: number analyzed (Participants) | 53
  Core Week 13 n=53 | 11.9 (10.98)
  Core Week 17 n=58: number analyzed (Participants) | 58
  Core Week 17 n=58 | 12.3 (9.03)
  Core Week 22 n=49: number analyzed (Participants) | 49
  Core Week 22 n=49 | 13.7 (13.82)
  Core Week 26 n=55: number analyzed (Participants) | 55
  Core Week 26 n=55 | 12.4 (12.09)
  Core Week 31 n=49: number analyzed (Participants) | 49
  Core Week 31 n=49 | 12.1 (11.02)
  Core Week 35 n=40: number analyzed (Participants) | 40
  Core Week 35 n=40 | 11.0 (8.71)
  Ext Week 43 n=23: number analyzed (Participants) | 23
  Ext Week 43 n=23 | 11.5 (8.12)
  Ext Week 51 n=21: number analyzed (Participants) | 21
  Ext Week 51 n=21 | 10.4 (6.80)
  Ext Week 59 n=23: number analyzed (Participants) | 23
  Ext Week 59 n=23 | 10.7 (6.89)
  Ext Week 67 n=22: number analyzed (Participants) | 22
  Ext Week 67 n=22 | 11.0 (7.23)
  Ext Week 75 n=22: number analyzed (Participants) | 22
  Ext Week 75 n=22 | 9.1 (4.16)
  Ext Week 83 n=19: number analyzed (Participants) | 19
  Ext Week 83 n=19 | 9.8 (8.20)
  Ext Week 91 n=19: number analyzed (Participants) | 19
  Ext Week 91 n=19 | 10.6 (8.34)
  Ext Week 99 n=16: number analyzed (Participants) | 16
  Ext Week 99 n=16 | 11.3 (8.50)
  Ext Week 107 n=13: number analyzed (Participants) | 13
  Ext Week 107 n=13 | 9.3 (6.61)
  Ext Week 115 n=15: number analyzed (Participants) | 15
  Ext Week 115 n=15 | 9.5 (7.22)
  Ext Week 123 n=14: number analyzed (Participants) | 14
  Ext Week 123 n=14 | 10.6 (8.24)
  Ext Week 131 n=12: number analyzed (Participants) | 12
  Ext Week 131 n=12 | 8.2 (6.01)
  Ext Week 139 n=10: number analyzed (Participants) | 10
  Ext Week 139 n=10 | 10.0 (7.01)
  Ext Week 147 n=9: number analyzed (Participants) | 9
  Ext Week 147 n=9 | 10.4 (7.02)
  Ext Week 155 n=9: number analyzed (Participants) | 9
  Ext Week 155 n=9 | 10.4 (7.02)
  Ext Week 163 n=5: number analyzed (Participants) | 5
  Ext Week 163 n=5 | 10.0 (4.85)
  Ext Week 171 n=5: number analyzed (Participants) | 5
  Ext Week 171 n=5 | 7.4 (3.36)
  Ext Week 179 n=5: number analyzed (Participants) | 5
  Ext Week 179 n=5 | 7.0 (3.32)
  Ext Week 187 n=5: number analyzed (Participants) | 5
  Ext Week 187 n=5 | 8.6 (5.32)
  Ext Week 195 n=4: number analyzed (Participants) | 4
  Ext Week 195 n=4 | 9.0 (4.76)
  Ext Week 203 n=4: number analyzed (Participants) | 4
  Ext Week 203 n=4 | 8.0 (2.94)
  Ext Week 211 n=3: number analyzed (Participants) | 3
  Ext Week 211 n=3 | 11.0 (4.58)
  Ext Week 219 n=2: number analyzed (Participants) | 2
  Ext Week 219 n=2 | 6.0 (0.00)
  Ext Week 227 n=2: number analyzed (Participants) | 2
  Ext Week 227 n=2 | 7.0 (1.41)
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 10.3 (3.21)
  Ext Week 243 n=1: number analyzed (Participants) | 1
  Ext Week 243 n=1 | 6.0
  Ext Week 251 n=1: number analyzed (Participants) | 1
  Ext Week 251 n=1 | 7.0
  Ext Week 267 n=1: number analyzed (Participants) | 1
  Ext Week 267 n=1 | 4.0

7. Secondary Outcome: Serum Cortisol Levels
Description: A pre-dose blood draw for an 8 am fasting serum cortisol measurement were taken at visits. Samples were analyzed by a central laboratory.
Time Frame: Baseline, weeks 2, 4, every 4 or 5 weeks during core, every 8 weeks during extension
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | All Patients
Number analyzed (Participants) | 68
nmol/L
  Baseline | 738.6 (332.53)
  Core Week 2 n-62: number analyzed (Participants) | 62
  Core Week 2 n-62 | 626.1 (281.57)
  Core Week 4 n=64: number analyzed (Participants) | 64
  Core Week 4 n=64 | 663.6 (292.38)
  Core Week 8 n=61: number analyzed (Participants) | 61
  Core Week 8 n=61 | 649.0 (297.11)
  Core Week 13 n=53: number analyzed (Participants) | 53
  Core Week 13 n=53 | 628.8 (269.43)
  Core Week 17 n=58: number analyzed (Participants) | 58
  Core Week 17 n=58 | 683.0 (282.28)
  Core Week 22 n=49: number analyzed (Participants) | 49
  Core Week 22 n=49 | 625.4 (216.29)
  Core Week 26 n=55: number analyzed (Participants) | 55
  Core Week 26 n=55 | 632.7 (278.75)
  Core Week 31 n=49: number analyzed (Participants) | 49
  Core Week 31 n=49 | 597.5 (247.60)
  Core Week 35 n=40: number analyzed (Participants) | 40
  Core Week 35 n=40 | 538.2 (205.40)
  Ext Week 43 n=23: number analyzed (Participants) | 23
  Ext Week 43 n=23 | 525.5 (178.63)
  Ext Week 51 n=21: number analyzed (Participants) | 21
  Ext Week 51 n=21 | 512.2 (243.59)
  Ext Week 59 n=21: number analyzed (Participants) | 21
  Ext Week 59 n=21 | 547.5 (193.67)
  Ext Week 67 n=22: number analyzed (Participants) | 22
  Ext Week 67 n=22 | 495.4 (213.03)
  Ext Week 75 n=21: number analyzed (Participants) | 21
  Ext Week 75 n=21 | 458.5 (170.88)
  Ext Week 83 n=19: number analyzed (Participants) | 19
  Ext Week 83 n=19 | 419.5 (141.26)
  Ext Week 91 n=19: number analyzed (Participants) | 19
  Ext Week 91 n=19 | 501.2 (235.89)
  Ext Week 99 n=16: number analyzed (Participants) | 16
  Ext Week 99 n=16 | 470.9 (248.0)
  Ext Week 107 n=13: number analyzed (Participants) | 13
  Ext Week 107 n=13 | 463.4 (189.27)
  Ext Week 115 n=15: number analyzed (Participants) | 15
  Ext Week 115 n=15 | 501.7 (212.27)
  Ext Week 123 n=14: number analyzed (Participants) | 14
  Ext Week 123 n=14 | 441.6 (150.98)
  Ext Week 131 n=12: number analyzed (Participants) | 12
  Ext Week 131 n=12 | 413.8 (325.5)
  Ext Week 139 n=10: number analyzed (Participants) | 10
  Ext Week 139 n=10 | 404.0 (90.87)
  Ext Week 147 n=10: number analyzed (Participants) | 10
  Ext Week 147 n=10 | 585.4 (216.92)
  Ext Week 155 n=8: number analyzed (Participants) | 8
  Ext Week 155 n=8 | 472.5 (122.96)
  Ext Week 163 n=6: number analyzed (Participants) | 6
  Ext Week 163 n=6 | 617.0 (212.11)
  Ext Week 171 n=5: number analyzed (Participants) | 5
  Ext Week 171 n=5 | 648.6 (243.79)
  Ext Week 179 n=5: number analyzed (Participants) | 5
  Ext Week 179 n=5 | 599.0 (388.78)
  Ext Week 187 n=5: number analyzed (Participants) | 5
  Ext Week 187 n=5 | 609.8 (292.85)
  Ext Week 195 n=4: number analyzed (Participants) | 4
  Ext Week 195 n=4 | 418.8 (138.69)
  Ext Week 203 n=4: number analyzed (Participants) | 4
  Ext Week 203 n=4 | 514.0 (212.27)
  Ext Week 211 n=3: number analyzed (Participants) | 3
  Ext Week 211 n=3 | 551.3 (339.87)
  Ext Week 219 n=2: number analyzed (Participants) | 2
  Ext Week 219 n=2 | 482.0 (25.46)
  Ext Week 227 n=2: number analyzed (Participants) | 2
  Ext Week 227 n=2 | 324.5 (177.48)
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 384.7 (165.17)
  Ext Week 243 n=1: number analyzed (Participants) | 1
  Ext Week 243 n=1 | 679.0
  Ext Week 251 n=1: number analyzed (Participants) | 1
  Ext Week 251 n=1 | 574.0
  Ext Week 267 n=1: number analyzed (Participants) | 1
  Ext Week 267 n=1 | 638.0

8. Secondary Outcome: Sitting Systolic Blood Pressure at Week 35
Description: The mean arterial blood pressure determinations were obtained in the sitting position. Three measurements were taken with 5 minute intervals and the mean was used for study specific procedures
Time Frame: Baseline and week 35
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 68
mmHg
  Baseline | 125.9 (14.3)
  Week 35 n=41: number analyzed (Participants) | 41
  Week 35 n=41 | 119.5 (18.6)

9. Secondary Outcome: Sitting Diastolic Blood Pressure at Week 35
Description: as for outcome 8
Time Frame: Baseline and week 35
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Patients
Number analyzed (Participants) | 68
mmHg
  Baseline | 81.8 (9.12)
  Week 35 n=41: number analyzed (Participants) | 41
  Week 35 n=41 | 77.2 (12.42)

10. Secondary Outcome: Body Weight at Week 35
Description: Weight was was one of the measures of clinical symptoms of CD
Time Frame: Baseline and week 35
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | All Patients
Number analyzed (Participants) | 68
kg
  Baseline | 82.2 (19.1)
  Week 35 n=41: number analyzed (Participants) | 41
  Week 35 n=41 | 75.6 (20.4)

11. Secondary Outcome: Body Mass Index at Week 35
Description: Body mass index was one of the measurements of clinical symptoms of CD. Body mass index=weight in kg divided by the square of the body height (in meters)
Time Frame: Baseline and week 35
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | All Patients
Number analyzed (Participants) | 68
kg/m2
  Baseline | 31.3 (6.6)
  Week 35 n=41: number analyzed (Participants) | 41
  Week 35 n=41 | 28.4 (6.8)

12. Secondary Outcome: Waist Circumference at Week 35
Description: Waist circumference was one of the measurements of clinical signs of CD
Time Frame: Baseline and week 35
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | All Patients
Number analyzed (Participants) | 68
cm
  Baseline | 104.1 (19.1)
  Week 35 n=41: number analyzed (Participants) | 41
  Week 35 n=41 | 99.1 (18.2)

13. Secondary Outcome: LDL, HDL and Total Cholesterol at Week 35
Description: LDL=Low density lipoprotein, HDL=high density llipoprotein and total protein were analyzed by a central laboratory
Time Frame: Baseline and week 35
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | All Patients
Number analyzed (Participants) | 68
mmol/L
  HDL Baseline | 1.5 (0.3)
  HDL Week 35 n=41: number analyzed (Participants) | 41
  HDL Week 35 n=41 | 1.5 (0.4)
  LDL Baseline | 3.2 (1.0)
  LDL Week 35 n=41: number analyzed (Participants) | 41
  LDL Week 35 n=41 | 2.8 (1.0)
  Total Baseline | 69.4 (3.7)
  Total Week 35 n=41: number analyzed (Participants) | 41
  Total Week 35 n=41 | 68.6 (4.8)

14. Secondary Outcome: Mean Scores of Cushing QoL Standardized Score at Week 17 and 35
Description: Patients who completed nine or more items for the 12-item Cushing's syndrome QoL questionaire were considered evaluable for that assessment. Raw scores were obtained for the 12 items using the following scoring: 1) always or very much, 2) often or quite a bit, 3) sometimes or somewhat, 4) rarely or very little, 5) never or not at all. Then the standardized score, Y, was calculated for each patient as follows: Y = 100* (X - n) / n*5 - n*1) = 100 * (X - n) / 4*n where X denoted the raw score and n the number of questions answered by the patient. The higher the score, the better the QoL. The best possible standardized score was 100 and the worst possible standardized score was 0
Time Frame: Baseline and week 17 and 35
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 68
scores on a scale
  Baseline Mean | 41.6 (20.2)
  Week 17 n=54: number analyzed (Participants) | 54
  Week 17 n=54 | 46.3 (19.7)
  Week 35 n=40: number analyzed (Participants) | 40
  Week 35 n=40 | 47.6 (20.8)

15. Secondary Outcome: Mean Scores of SF-12v2 Domain Scores at Week 17 and 35
Description: SF-12v2 General Health Survey is a general patient reported outcome instrument over time. It is scored to provide eight health domain scores (Bodily Pain (BP), General Health (GH), Physical Functioning (PF), Role-Physical (RP), Social Functioning (SF), Role-Emotional (RE), Vitality (VT) and Mental Health (MH)). These eight domain scores can be combined to form two summary scores reflecting overall physical and mental health: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The analyses reported here focus on PCS and MCS scores. The domain scores use a norm-based score, which standardizes the scores with respect to the mean and standard deviation of a nationally representative sample of United States (US) adults. These are the scores on the original scale which have not been transformed in any way. The possible range of scores is 0 to 100, with higher scores representing better outcomes.
Time Frame: Baseline, week 17 and 35
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 68
scores on a scale
  Baseline Bodily pain scale | 42.9 (11.93)
  Week 17 n=52 Bodily pain scale: number analyzed (Participants) | 52
  Week 17 n=52 Bodily pain scale | 45.1 (10.75)
  Week 35 n=40 Bodily pain scale: number analyzed (Participants) | 40
  Week 35 n=40 Bodily pain scale | 44.9 (10.79)
  Baseline n=67 General health scale:: number analyzed (Participants) | 67
  Baseline n=67 General health scale: | 38.9 (9.23)
  Week 17 n=52 General health scale:: number analyzed (Participants) | 52
  Week 17 n=52 General health scale: | 40.9 (8.52)
  Week 35 n=40 General health scale:: number analyzed (Participants) | 40
  Week 35 n=40 General health scale: | 40.7 (8.94)
  Baseline n=67 Mental component: number analyzed (Participants) | 67
  Baseline n=67 Mental component | 42.4 (10.17)
  Week 17 n=52 Mental component: number analyzed (Participants) | 52
  Week 17 n=52 Mental component | 41.9 (9.68)
  Week 35 n=40 Mental component: number analyzed (Participants) | 40
  Week 35 n=40 Mental component | 42.1 (8.32)
  Baseline n=67 Mental health: number analyzed (Participants) | 67
  Baseline n=67 Mental health | 41.9 (10.48)
  Week 17 n=52 Mental health: number analyzed (Participants) | 52
  Week 17 n=52 Mental health | 43.0 (9.54)
  Week 35 n=40 Mental health: number analyzed (Participants) | 40
  Week 35 n=40 Mental health | 42.4 (8.44)
  Baseline n=67 Physical component summary: number analyzed (Participants) | 67
  Baseline n=67 Physical component summary | 42.7 (9.03)
  Week 17 n=52 Physical component summary: number analyzed (Participants) | 52
  Week 17 n=52 Physical component summary | 44.0 (8.52)
  Week 35 n=40 Physical component summary: number analyzed (Participants) | 40
  Week 35 n=40 Physical component summary | 43.4 (9.59)
  Baseline n=67 Physical functioning: number analyzed (Participants) | 67
  Baseline n=67 Physical functioning | 42.1 (10.17)
  Week 17 n=52 Physical functioning: number analyzed (Participants) | 52
  Week 17 n=52 Physical functioning | 41.9 (8.93)
  Week 35 n=40 Physical functioning: number analyzed (Participants) | 40
  Week 35 n=40 Physical functioning | 42.1 (11.10)
  Baseline n=67 Role emotional: number analyzed (Participants) | 67
  Baseline n=67 Role emotional | 39.7 (11.67)
  Week 17 n=52 Role emotional: number analyzed (Participants) | 52
  Week 17 n=52 Role emotional | 38.0 (9.95)
  Week 35 n=40 Role emotional: number analyzed (Participants) | 40
  Week 35 n=40 Role emotional | 38.7 (10.70)
  Baseline n=67 Role physical scale:: number analyzed (Participants) | 67
  Baseline n=67 Role physical scale: | 42.3 (10.45)
  Week 17 n=52 Role physical scale:: number analyzed (Participants) | 52
  Week 17 n=52 Role physical scale: | 42.8 (8.73)
  Week 35 n=40 Role physical scale:: number analyzed (Participants) | 40
  Week 35 n=40 Role physical scale: | 41.3 (9.63)
  Baseline n=67 Social functioning: number analyzed (Participants) | 67
  Baseline n=67 Social functioning | 42.2 (11.22)
  Week 17 n=52 Social functioning: number analyzed (Participants) | 52
  Week 17 n=52 Social functioning | 43.0 (8.70)
  Week 35 n=40 Social functioning: number analyzed (Participants) | 40
  Week 35 n=40 Social functioning | 43.3 (9.66)
  Baseline n=67 Vitality scale:: number analyzed (Participants) | 67
  Baseline n=67 Vitality scale: | 47.2 (10.02)
  Week 17 n=52 Vitality scale:: number analyzed (Participants) | 52
  Week 17 n=52 Vitality scale: | 45.7 (10.29)
  Week 35 n=40 Vitality scale:: number analyzed (Participants) | 40
  Week 35 n=40 Vitality scale: | 45.6 (8.78)

16. Secondary Outcome: Number of Participants With Improvement in Clinical Symptom of Hypercortisolism From Baseline - Facial Rubor
Description: Clinical symptoms include: facial rubor, hirsutism, striae, and supraclavicular and dorsal fat pad. Two photographs, one frontal and one lateral from the shoulders up were taken to assess facial plethora, supraclavicular and dorsal fat pads. Two photographs, frontal and dorsal of the trunk with patient in standing position were taken to assess striae, and hirsutism. The photographs were assessed by a qualified physician at the site. Improvement=decrease in severity of symptom since baseline
Time Frame: Baseline, weeks 2, 4, every 4 or 5 weeks during core, every 16 weeks during extension
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 68
participants
  Core Week 1 n=40: number analyzed (Participants) | 40
  Core Week 1 n=40 | 5
  Core Week 2 n=37: number analyzed (Participants) | 37
  Core Week 2 n=37 | 8
  Core Week 4 n=38: number analyzed (Participants) | 38
  Core Week 4 n=38 | 8
  Core Week 8 n=37: number analyzed (Participants) | 37
  Core Week 8 n=37 | 12
  Core Week 13 n=32: number analyzed (Participants) | 32
  Core Week 13 n=32 | 11
  Core Week 17 n=32: number analyzed (Participants) | 32
  Core Week 17 n=32 | 11
  Core Week 22 n=28: number analyzed (Participants) | 28
  Core Week 22 n=28 | 10
  Core Week 26 n=31: number analyzed (Participants) | 31
  Core Week 26 n=31 | 14
  Core Week 31 n=32: number analyzed (Participants) | 32
  Core Week 31 n=32 | 15
  Core Week 35 n=26: number analyzed (Participants) | 26
  Core Week 35 n=26 | 13
  Ext Week 43 n=11: number analyzed (Participants) | 11
  Ext Week 43 n=11 | 2
  Ext Week 59 n=11: number analyzed (Participants) | 11
  Ext Week 59 n=11 | 3
  Ext Week 75 n=12: number analyzed (Participants) | 12
  Ext Week 75 n=12 | 3
  Ext Week 91 n=10: number analyzed (Participants) | 10
  Ext Week 91 n=10 | 3
  Ext Week 107 n=9: number analyzed (Participants) | 9
  Ext Week 107 n=9 | 3
  Ext Week 123 n=10: number analyzed (Participants) | 10
  Ext Week 123 n=10 | 2
  Ext Week 139 n=7: number analyzed (Participants) | 7
  Ext Week 139 n=7 | 2
  Ext Week 155 n=4: number analyzed (Participants) | 4
  Ext Week 155 n=4 | 0
  Ext Week 171 n=3: number analyzed (Participants) | 3
  Ext Week 171 n=3 | 0
  Ext Week 187 n=3: number analyzed (Participants) | 3
  Ext Week 187 n=3 | 0
  Ext Week 203 n=4: number analyzed (Participants) | 4
  Ext Week 203 n=4 | 0
  Ext Week 219 n=2: number analyzed (Participants) | 2
  Ext Week 219 n=2 | 0
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 0
  Ext Week 251 n=1: number analyzed (Participants) | 1
  Ext Week 251 n=1 | 0
  Ext Week 267 n=1: number analyzed (Participants) | 1
  Ext Week 267 n=1 | 0

17. Secondary Outcome: Number of Participants With Improvement in Clinical Symptom of Hypercortisolism From Baseline - Hirsutism
Description: as for outcome 16
Time Frame: Baseline, weeks 2, 4, every 4 or 5 weeks during core, every 16 weeks during extension
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 68
participants
  Core Week 1 n=35: number analyzed (Participants) | 35
  Core Week 1 n=35 | 5
  Core Week 2 n-33: number analyzed (Participants) | 33
  Core Week 2 n-33 | 3
  Core Week 4 n=32: number analyzed (Participants) | 32
  Core Week 4 n=32 | 4
  Core Week 8 n=32: number analyzed (Participants) | 32
  Core Week 8 n=32 | 4
  Core Week 13 n=27: number analyzed (Participants) | 27
  Core Week 13 n=27 | 4
  Core Week 17 n=28: number analyzed (Participants) | 28
  Core Week 17 n=28 | 3
  Core Week 22 n=25: number analyzed (Participants) | 25
  Core Week 22 n=25 | 5
  Core Week 26 n=27: number analyzed (Participants) | 27
  Core Week 26 n=27 | 8
  Core Week 31 n=28: number analyzed (Participants) | 28
  Core Week 31 n=28 | 9
  Core Week 35 n=23: number analyzed (Participants) | 23
  Core Week 35 n=23 | 7
  Ext Week 43 n=10: number analyzed (Participants) | 10
  Ext Week 43 n=10 | 2
  Ext Week 59 n=9: number analyzed (Participants) | 9
  Ext Week 59 n=9 | 2
  Ext Week 75 n=10: number analyzed (Participants) | 10
  Ext Week 75 n=10 | 3
  Ext Week 91 n=9: number analyzed (Participants) | 9
  Ext Week 91 n=9 | 2
  Ext Week 107 n=8: number analyzed (Participants) | 8
  Ext Week 107 n=8 | 1
  Ext Week 123 n=9: number analyzed (Participants) | 9
  Ext Week 123 n=9 | 2
  Ext Week 139 n=7: number analyzed (Participants) | 7
  Ext Week 139 n=7 | 2
  Ext Week 155 n=4: number analyzed (Participants) | 4
  Ext Week 155 n=4 | 2
  Ext Week 171 n=4: number analyzed (Participants) | 4
  Ext Week 171 n=4 | 2
  Ext Week 187 n=3: number analyzed (Participants) | 3
  Ext Week 187 n=3 | 2
  Ext Week 203 n=4: number analyzed (Participants) | 4
  Ext Week 203 n=4 | 2
  Ext Week 219 n=2: number analyzed (Participants) | 2
  Ext Week 219 n=2 | 1
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 1
  Ext Week 251 n=1: number analyzed (Participants) | 1
  Ext Week 251 n=1 | 0
  Ext Week 267 n=1: number analyzed (Participants) | 1
  Ext Week 267 n=1 | 0

18. Secondary Outcome: Number of Participants With Improvement in Clinical Symptom of Hypercortisolism From Baseline - Striae
Description: as for outcome 16
Time Frame: Baseline, weeks 2, 4, every 4 or 5 weeks during core, every 16 weeks during extension
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 68
participants
  Core Week 1 n=40: number analyzed (Participants) | 40
  Core Week 1 n=40 | 5
  Core Week 2 n-37: number analyzed (Participants) | 37
  Core Week 2 n-37 | 2
  Core Week 4 n=38: number analyzed (Participants) | 38
  Core Week 4 n=38 | 5
  Core Week 8 n=37: number analyzed (Participants) | 37
  Core Week 8 n=37 | 8
  Core Week 13 n=32: number analyzed (Participants) | 32
  Core Week 13 n=32 | 7
  Core Week 17 n=32: number analyzed (Participants) | 32
  Core Week 17 n=32 | 7
  Core Week 22 n=28: number analyzed (Participants) | 28
  Core Week 22 n=28 | 7
  Core Week 26 n=31: number analyzed (Participants) | 31
  Core Week 26 n=31 | 9
  Core Week 31 n=32: number analyzed (Participants) | 32
  Core Week 31 n=32 | 12
  Core Week 35 n=26: number analyzed (Participants) | 26
  Core Week 35 n=26 | 8
  Ext Week 43 n11=: number analyzed (Participants) | 11
  Ext Week 43 n11= | 1
  Ext Week 59 n=11: number analyzed (Participants) | 11
  Ext Week 59 n=11 | 1
  Ext Week 75 n=12: number analyzed (Participants) | 12
  Ext Week 75 n=12 | 1
  Ext Week 91 n=10: number analyzed (Participants) | 10
  Ext Week 91 n=10 | 1
  Ext Week 107 n=9: number analyzed (Participants) | 9
  Ext Week 107 n=9 | 0
  Ext Week 123 n=10: number analyzed (Participants) | 10
  Ext Week 123 n=10 | 0
  Ext Week 139 n=7: number analyzed (Participants) | 7
  Ext Week 139 n=7 | 0
  Ext Week 155 n=4: number analyzed (Participants) | 4
  Ext Week 155 n=4 | 1
  Ext Week 171 n=3: number analyzed (Participants) | 3
  Ext Week 171 n=3 | 0
  Ext Week 187 n=3: number analyzed (Participants) | 3
  Ext Week 187 n=3 | 0
  Ext Week 203 n=4: number analyzed (Participants) | 4
  Ext Week 203 n=4 | 1
  Ext Week 219 n=2: number analyzed (Participants) | 2
  Ext Week 219 n=2 | 0
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 1
  Ext Week 251 n=1: number analyzed (Participants) | 1
  Ext Week 251 n=1 | 0
  Ext Week 267 n=1: number analyzed (Participants) | 1
  Ext Week 267 n=1 | 1

19. Secondary Outcome: Number of Participants With Improvement in Clinical Symptom of Hypercortisolism From Baseline - Supraclavicular Fat Pad
Description: as for outcome 16
Time Frame: Baseline, weeks 2, 4, every 4 or 5 weeks during core, every 8 weeks during extension
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 68
participants
  Core Week 1 n=40: number analyzed (Participants) | 40
  Core Week 1 n=40 | 6
  Core Week 2 n-37: number analyzed (Participants) | 37
  Core Week 2 n-37 | 7
  Core Week 4 n=37: number analyzed (Participants) | 37
  Core Week 4 n=37 | 6
  Core Week 8 n=37: number analyzed (Participants) | 37
  Core Week 8 n=37 | 8
  Core Week 13 n=32: number analyzed (Participants) | 32
  Core Week 13 n=32 | 8
  Core Week 17 n=32: number analyzed (Participants) | 32
  Core Week 17 n=32 | 9
  Core Week 22 n=28: number analyzed (Participants) | 28
  Core Week 22 n=28 | 9
  Core Week 26 n=31: number analyzed (Participants) | 31
  Core Week 26 n=31 | 10
  Core Week 31 n=32: number analyzed (Participants) | 32
  Core Week 31 n=32 | 12
  Core Week 35 n=26: number analyzed (Participants) | 26
  Core Week 35 n=26 | 11
  Ext Week 43 n=11: number analyzed (Participants) | 11
  Ext Week 43 n=11 | 1
  Ext Week 59 n=11: number analyzed (Participants) | 11
  Ext Week 59 n=11 | 0
  Ext Week 75 n=12: number analyzed (Participants) | 12
  Ext Week 75 n=12 | 1
  Ext Week 91 n=10: number analyzed (Participants) | 10
  Ext Week 91 n=10 | 1
  Ext Week 107 n=9: number analyzed (Participants) | 9
  Ext Week 107 n=9 | 0
  Ext Week 123 n=10: number analyzed (Participants) | 10
  Ext Week 123 n=10 | 1
  Ext Week 139 n=7: number analyzed (Participants) | 7
  Ext Week 139 n=7 | 1
  Ext Week 155 n=4: number analyzed (Participants) | 4
  Ext Week 155 n=4 | 1
  Ext Week 171 n=3: number analyzed (Participants) | 3
  Ext Week 171 n=3 | 1
  Ext Week 187 n=3: number analyzed (Participants) | 3
  Ext Week 187 n=3 | 1
  Ext Week 203 n=4: number analyzed (Participants) | 4
  Ext Week 203 n=4 | 1
  Ext Week 219 n=2: number analyzed (Participants) | 2
  Ext Week 219 n=2 | 1
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 2
  Ext Week 251 n=1: number analyzed (Participants) | 1
  Ext Week 251 n=1 | 0
  Ext Week 267 n=1: number analyzed (Participants) | 1
  Ext Week 267 n=1 | 0

20. Secondary Outcome: Number of Participants With Improvement in Clinical Symptom of Hypercortisolism From Baseline - Dorsal Fat Pad
Description: as for outcome 16
Time Frame: Baseline, weeks 2, 4, every 4 or 5 weeks during core, every 16 weeks during extension
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 68
participants
  Core Week 1 n=40: number analyzed (Participants) | 40
  Core Week 1 n=40 | 6
  Core Week 2 n-37: number analyzed (Participants) | 37
  Core Week 2 n-37 | 4
  Core Week 4 n=37: number analyzed (Participants) | 37
  Core Week 4 n=37 | 5
  Core Week 8 n=37: number analyzed (Participants) | 37
  Core Week 8 n=37 | 5
  Core Week 13 n=32: number analyzed (Participants) | 32
  Core Week 13 n=32 | 4
  Core Week 17 n=32: number analyzed (Participants) | 32
  Core Week 17 n=32 | 8
  Core Week 22 n=28: number analyzed (Participants) | 28
  Core Week 22 n=28 | 8
  Core Week 26 n=31: number analyzed (Participants) | 31
  Core Week 26 n=31 | 12
  Core Week 31 n=32: number analyzed (Participants) | 32
  Core Week 31 n=32 | 13
  Core Week 35 n=26: number analyzed (Participants) | 26
  Core Week 35 n=26 | 9
  Ext Week 43 n=11: number analyzed (Participants) | 11
  Ext Week 43 n=11 | 3
  Ext Week 59 n=10: number analyzed (Participants) | 10
  Ext Week 59 n=10 | 4
  Ext Week 75 n=12: number analyzed (Participants) | 12
  Ext Week 75 n=12 | 5
  Ext Week 91 n=10: number analyzed (Participants) | 10
  Ext Week 91 n=10 | 3
  Ext Week 107 n=9: number analyzed (Participants) | 9
  Ext Week 107 n=9 | 2
  Ext Week 123 n=10: number analyzed (Participants) | 10
  Ext Week 123 n=10 | 3
  Ext Week 139 n=7: number analyzed (Participants) | 7
  Ext Week 139 n=7 | 3
  Ext Week 155 n=4: number analyzed (Participants) | 4
  Ext Week 155 n=4 | 1
  Ext Week 171 n=3: number analyzed (Participants) | 3
  Ext Week 171 n=3 | 1
  Ext Week 187 n=3: number analyzed (Participants) | 3
  Ext Week 187 n=3 | 2
  Ext Week 203 n=4: number analyzed (Participants) | 4
  Ext Week 203 n=4 | 1
  Ext Week 219 n=2: number analyzed (Participants) | 2
  Ext Week 219 n=2 | 1
  Ext Week 235 n=3: number analyzed (Participants) | 3
  Ext Week 235 n=3 | 2
  Ext Week 251 n=1: number analyzed (Participants) | 1
  Ext Week 251 n=1 | 0
  Ext Week 267 n=1: number analyzed (Participants) | 1
  Ext Week 267 n=1 | 0

21. Secondary Outcome: Number of Participants With Shift From Mild to Severe in Clinical Signs of Hypercortisolism
Description: Facial rubor, hirsutism, striae, and supraclavicular and dorsal fat pad were assessed. Two photographs, one frontal and one lateral from the shoulders up will be taken to assess facial plethora, supraclavicular and dorsal fat pads. Two photographs, frontal and dorsal of the trunk with patient in standing position will be taken to assess striae, and hirsutism. The photographs must be assessed by a qualified physician at the site. Improvement=decrease in severity of symptom since baseline
Time Frame: Baseline, weeks 1, 2, 4, every 4 or 5 weeks during core, every 8 weeks during extension
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 68
participants
  Core Week 4 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Core Week 4 Facial rubor baseline n=17 | 1
  Core Week 35 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Core Week 35 Facial rubor baseline n=17 | 1
  Ext Week 43 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Ext Week 43 Facial rubor baseline n=17 | 1
  Ext Week 59 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Ext Week 59 Facial rubor baseline n=17 | 1
  Ext Week 67 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Ext Week 67 Facial rubor baseline n=17 | 1
  Ext Week 83 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Ext Week 83 Facial rubor baseline n=17 | 1
  Ext Week 91 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Ext Week 91 Facial rubor baseline n=17 | 1
  Ext Week 99 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Ext Week 99 Facial rubor baseline n=17 | 1
  Ext Week 107 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Ext Week 107 Facial rubor baseline n=17 | 1
  Ext Week 115 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Ext Week 115 Facial rubor baseline n=17 | 1
  Ext Week 123 Facial rubor baseline n=17: number analyzed (Participants) | 17
  Ext Week 123 Facial rubor baseline n=17 | 1
  Core Week 1 Hirsutism baseline n=12: number analyzed (Participants) | 12
  Core Week 1 Hirsutism baseline n=12 | 1
  Core Week 2 Hirsutism baseline n=12: number analyzed (Participants) | 12
  Core Week 2 Hirsutism baseline n=12 | 1
  Ext Week 59 Striae baseline n=10: number analyzed (Participants) | 10
  Ext Week 59 Striae baseline n=10 | 1
  Ext Week 99 Striae baseline n=10: number analyzed (Participants) | 10
  Ext Week 99 Striae baseline n=10 | 1
  Ext Week 107 Striae baseline n=10: number analyzed (Participants) | 10
  Ext Week 107 Striae baseline n=10 | 1
  Ext Week 115 Striae baseline n=10: number analyzed (Participants) | 10
  Ext Week 115 Striae baseline n=10 | 1
  Ext Week 123 Striae baseline n=10: number analyzed (Participants) | 10
  Ext Week 123 Striae baseline n=10 | 1
  Ext Week 99 Supraclavicular fat pad BL n=17: number analyzed (Participants) | 17
  Ext Week 99 Supraclavicular fat pad BL n=17 | 1
  Ext Week 107 Supraclavicular fat pad BL n=17: number analyzed (Participants) | 17
  Ext Week 107 Supraclavicular fat pad BL n=17 | 1

22. Secondary Outcome: Number of Patients With Shift From Standing Easily to Not Being Able to Stand
Description: To test proximal muscle strength patients should be placed in a low seated position (for instance on an examination room stool). They should be asked to extend the arms in front of them. From this seated position patients will be asked to stand up. Patients will be evaluated using the following scale: 3. - completely unable to stand 2. - able to stand only by using arms as assistance
  1. - able to stand after several efforts without using arms as assistance 0. - able to stand easily with arms extended
Time Frame: Baseline up to week 267
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 68
participants
  Core Week 26: number analyzed (Participants) | 41
  Core Week 26 | 1
  Core Week 35: number analyzed (Participants) | 32
  Core Week 35 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 28 days post treatment, up to maximum duration of 272 weeks
Description: Any sign or symptom that occurs during the study treatment plus 28 days post treatment
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 3/68
Serious Adverse Events (participants affected / at risk) | 15/68
Other Adverse Events (participants affected / at risk) | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=68)
Anaemia (Blood and lymphatic system disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Glucocorticoid deficiency (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Intra-abdominal haematoma (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Abscess limb (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=68)
Anaemia (Blood and lymphatic system disorders) | 6
Bradycardia (Cardiac disorders) | 4
Mitral valve incompetence (Cardiac disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 30
Flatulence (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 35
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 7
Fatigue (General disorders) | 13
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 4
Cholelithiasis (Hepatobiliary disorders) | 22
Hepatic steatosis (Hepatobiliary disorders) | 4
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 6
Alanine aminotransferase increased (Investigations) | 5
Gamma-glutamyltransferase increased (Investigations) | 11
Decreased appetite (Metabolism and nutrition disorders) | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 12
Glucose tolerance impaired (Metabolism and nutrition disorders) | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 35
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 11
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 13
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 19
Headache (Nervous system disorders) | 20
Somnolence (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 4
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 8
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT01915303/SAP_000.pdf
  • Study Protocol (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT01915303/Prot_001.pdf